CLINICAL TRIAL: NCT06212323
Title: Smoldering Myeloma High-Risk Patient Observation and Longitudinal Insight Trial
Acronym: SPOTLIGHT
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: HCI170107
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Smoldering Multiple Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients with smoldering myeloma undergoing active surveillance with diffusion weighted whole body MRI. — Patients with high-risk smoldering myeloma will be prospectively followed and chart review will be performed to determine if progression events happen, and how they happen.
  All patients on the study are recommended to undergo the following standard of care surveillance protocol:
  * Complete Blood Count (CBC), Complete Metabolic Panel (CMP), myeloma blood tests (serum kappa/lambda light chains, monoclonal protein evaluation, immunoglobulin levels), to be done monthly for first year, and then every two months for the second year.
  * WB DW-MRIs every 6 months during the study period.
  * 24-hour urine Immunofixation/electrophoresis is expected to be completed approximately every 6 months.
  * Bone marrow biopsy will be performed annually during the study time-period.

SUMMARY:
The purpose of this study is to define the natural history of high-risk smoldering myeloma in a modern cohort of patients undergoing close standard of care follow-up with diffusion weighted whole body magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject aged ≥ 18 years.
* Diagnosis of smoldering myeloma as per the IMWG criteria, specifically:

  * Serum monoclonal protein (IgG or IgA) of 30g/L or greater per 24 hours or urinary monoclonal protein of 500mg or greater per 24 hours and/or
  * Clonal bone marrow plasma cells 10-59% with the absence of myeloma-defining events or amyloidosis
* High-risk smoldering myeloma defined as two or more out of four of the following criteria:

  * M-spike greater than 2 g/dL
  * An involved/uninvolved free light chain ratio greater than 20
  * Bone marrow plasmacytosis greater than 20%
  * Presence of any of translocation (4;14), deletion 17p, deletion 13q or 1q gain by conventional cytogenetics/fluorescence in situ hybridization (FISH) studies) and/or
  * An IMWG SMM score of 9 or greater according to the IMWG risk model for smoldering multiple myeloma (SMM)
* Diagnosis of high-risk SMM made within 365 days of enrollment in the study. Note: If a patient previously had MGUS or low/intermediate SMM- the date at which high-risk SMM was diagnosed would have to be within 365 days of enrollment in the study.

Exclusion Criteria:

* Presence of any features that would meet diagnostic criteria for myeloma as per the IMWG Criteria
* Presence of extramedullary plasmacytomas
* Presence of any focal bone marrow lesions, or lytic bone lesions on imaging done prior to screening or on screening. However, presence of diffuse or patchy infiltration of the marrow (without any clear lesions) on MRI, will not be an exclusion criteria. Patients with 1 focal marrow lesion on MRI that is attributable to plasma cell dyscrasia, will be excluded from study, even if they do not meet criteria for myeloma.
* Creatinine clearance of less than 40ml/min.
* Presence of AL Amyloidosis (the amount of workup necessary to exclude AL Amyloidosis is per the discretion of the treating investigator, however the investigator must attest that they do not believe AL Amyloidosis to be present at time of enrollment. Serum nt-PROBNP is recommended as part of evaluation in order to ascertain for cardiac amyloidosis).
* Hemoglobin of less than 11g/dl, unless a clearly reversible reason for anemia is identified, at which point they can be rescreened in two months if Hgb is greater than 11g/dl.

Note: The Hgb cut-offs can vary between institutions (lower cut-off for Hgb University of Utah for men is a Hgb of 14.8, rendering a patient with Hgb of 12.7 as having a CRAB feature). If the Hgb is above 10g/dl but the patient meets the definition of anemia according to the IMWG criteria, by virtue of this being more than 2 g/dl below the limit of normal, the investigator can decide whether to call a patient being considered for screening as having multiple myeloma OR smoldering myeloma and allow enrollment on this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Smoldering myeloma (SMM)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of morbid progression events attributable to a plasma cell dyscrasia at two years, with morbid events defined as: death, renal injury that does not reverse, fracture, lytic bone lesion, AL Amyloidosis or plasma cell leukemia. | 2 years
  Frequency and nature of progression events in a prospective cohort of patients with smoldering myeloma undergoing active surveillance with diffusion weighted whole body MRI

SECONDARY OUTCOMES:
Change in the quality of life as measured by physical function domain on the PROMIS-29 (Patient-Reported Outcomes Measurement Information System), from baseline to the end of study at 24 months of follow-up. | 2 years
  Determine longitudinal Quality of Life as assessed by the PROMIS-29 instrument. The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of physical function.
Change in the quality of life as measured by pain interference domain on the PROMIS-29 (Patient-Reported Outcomes Measurement Information System), from baseline to the end of study at 24 months of follow-up. | 2 years
  Determine longitudinal Quality of Life as assessed by the PROMIS-29 instrument. The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of pain interference.
Change in the quality of life as measured by anxiety domain on the PROMIS-29 (Patient-Reported Outcomes Measurement Information System), from baseline to the end of study at 24 months of follow-up. | 2 years
  Determine longitudinal Quality of Life as assessed by the PROMIS-29 instrument. The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Rehman Mohyuddin, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT06212323/Prot_SAP_000.pdf